CLINICAL TRIAL: NCT03536845
Title: Vitamin D Supplementation to Prevent Vitamin D Deficiency for Children With Epilepsy: a Randomized Controlled Clinical Trial
Brief Title: Vitamin D Supplementation to Prevent Vitamin D Deficiency for Children With Epilepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: King Saud University (Other)
Collaborators: Dallah hospital (Unknown)
Responsible Party: Principal Investigator, Reem Al Khalifah, Assistant Professor, King Saud University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: E-17-2425
Record Dates: First submitted 2018-05-14; First posted 2018-05-25 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Epilepsy; Vitamin D Deficiency
MeSH Terms: conditions — Epilepsy; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 400 IU (Active Comparator)
  Interventions: Drug: Vitamin D 3
- 1000 IU (Active Comparator)
  Interventions: Drug: Vitamin D 3

INTERVENTIONS:
Drug: Vitamin D 3 — oral drops

SUMMARY:
To determine the maintenance dose of vitamin D supplementation required for children with epilepsy to maintain normal vitamin D level.

DETAILED DESCRIPTION:
children aged 2-16 years diagnosed with idiopathic epilepsy will be randomized to receive either cholecalciferol doses (400IU vs 1000IU) with follow up at 3 and 6 months post supplementation.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged between 2-16 years who were diagnosed with Epilepsy and being treated with AEDs
2. Followed up in the outpatient pediatric neurology clinic at King Khalid University Hospital during the period of two years.

Exclusion Criteria:

1. Children with pre-existing vitamin D metabolism problems; because they are known to need different vitamin D doses and monitoring for clinical improvement:

   * Vitamin D dependent rickets
   * Malabsorption syndromes like celiac disease, inflammatory bowel disease
   * Renal disease
   * Hepatic disease
2. Children who are not safe to start vitamin D supplementation; because vitamin D supplementation will causes toxicity and induces nephrocalcinosis:

   * Hypercalcemia at baseline total corrected calcium >2.5mg/dl
   * Vitamin D level > 250 nmol/L
   * Urine calcium: creatinine ration > 1.2 mol/mol, or > 0.41g/g.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 116 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Vitamin D level < 75 nmol/L | 6 months of supplementation

SECONDARY OUTCOMES:
Seizure rate | 6 months of supplementation
bone mineral density (BMD) measurement | 6 months of supplementation
Cost- effectiveness of vitamin D supplementation | 6 months of supplementation
  cost of vitamin D supplementation compared to the cost of poor bone health, hospital admission
Safety: Prevalence of hypercalcemia total calcium >2.7mg/dl, 25 OH vit D level> 250 nmol/l, and Urine calcium: creatinine ration > 1.2 mol/mol, or > 0.41g/g. | 6 months of supplementation

OTHER OUTCOMES:
Vitamin D level < 75 nmol/L | 6 months of supplementation
  subgroup analysis among enzyme inducer and non-enzyme inducer (anti-epileptic medications) AEDs
Vitamin D level < 75 nmol/L | 6 months of supplementation
  subgroup analysis among obese and non-obese patients

CONTACTS AND LOCATIONS:
Overall Officials: Reem Al Khalifah, Principal Investigator — King Saud University
Locations (1):
- Reem ALKhalifah, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
URL: https://journals.lww.com/md-journal/Fulltext/2018/10050/Vitamin_D_supplementation_to_prevent_vitamin_D.99.aspx